CLINICAL TRIAL: NCT01362855
Title: Advance Care Planning Evaluation in Hospitalized Elderly Patients: A Multicenter, Prospective Study
Brief Title: Advance Care Planning Evaluation in Hospitalized Elderly Patients
Acronym: ACCEPT
Status: Completed | Type: Observational
Sponsor: Daren K. Heyland (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor-Investigator, Daren K. Heyland, Director, Clinical Evaluation Reserach Unit, Clinical Evaluation Research Unit at Kingston General Hospital
Organization: Clinical Evaluation Research Unit at Kingston General Hospital (Other)
Other Study IDs: ACCEPT Study
Record Dates: First submitted 2011-05-20; First posted 2011-05-30 (Estimated); Last update posted 2020-12-16 (Actual); Status verified 2015-02

CONDITIONS: Critical Illness; Chronic Obstructive Lung Disease; Congestive Heart Failure; Cirrhosis; Cancer
Keywords: Advance Care Planning; End of life; Knowledge translation; Goals of care; Advance directive; Living will
MeSH Terms: conditions — Critical Illness; Pulmonary Disease, Chronic Obstructive; Heart Failure; Fibrosis; Neoplasms; Death

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the study is to inform decision-makers of the best strategies to implement advanced care planning (ACP).

An advanced care plan (ACP) is a verbal or written instruction describing what kind of care an individual would want (or not want)if they are no longer able speak for themselves to make health care decisions.

DETAILED DESCRIPTION:
Advance Care Planning (ACP) may offer some assistance with reducing health care costs for older Canadians and yet, at the same time, improving quality of care. ACP is the process by which a person considers options about future health care decisions and identifies their wishes. ACP has been shown to increase the quality of life of dying patients, improve the experience of family members, and decrease health care costs.

There have been initiatives leading to the development and implementation of system-wide strategies to increase ACP, however there has been no evaluation of the effectiveness of these efforts from the perspective of patients and families. Many questions pertaining to barriers and facilitators to implementation and impact of ACP on outcomes in Canada remain.

The investigators propose to conduct a perspective audit of current practice related to ACP in elderly patients at high-risk for dying and their families. The investigators will determine the extent to which these patients and families have engaged in ACP, what barriers and facilitators they preceive, and how satisfied they are with communication and decision making at the end of life. Informed by a baseline evaluation of site strengths, weaknesses and barriers, the investigators propose to develop tailored interventions to enable participating sites to improve their success with ACP during the entire study period. By repeating the audit and feedback cycle annually, the investigators will enable sites to make continuous efforts to improve their performance and be able to evaluate the effect of our audit/feedback/tailored intervention strategy compared to baseline. Additionally, for those patients who have engaged in ACP activities, the investigators can compare their outcomes to those who have not.

The overall goal of this study is to inform decision-makers as the best strategies to implement advance care planning (ACP).

ELIGIBILITY:
Inclusion Criteria:

* 55 years or older with one or more of the following diagnoses:

  * Chronic obstructive lung disease - 2 of the 4 of: baseline PaCO2 of > 45 torr, cor pulmonale; respiratory failure episode within the preceding year; forced expiratory volume in 1 sec <0.5 L.
  * Congestive heart failure - New York Heart Association class IV symptoms and left ventricular ejection fraction < 25%.
  * Cirrhosis - confirmed by imaging studies or documentation of esophageal varices and one of three conditions: a) hepatic coma, b) Child's class C liver disease, or c) Child's class B liver disease with gastrointestinal bleeding.
  * Cancer - metastatic cancer or stage IV lymphoma.
  * End-stage dementia (inability to perform all ADLs, mutism or minimal verbal output secondary to dementia, bed-bound state prior to acute illness) OR
* Any patient 80 years of age or older admitted to hospital from the community because of an acute medical or surgical condition.

Exclusion Criteria:

* Non-English speaking patient/family member
* Patient with cognitive impairment

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We will enroll patients who are at high risk of dying and/or their families (where available).
Sampling Method: Probability Sample
Enrollment: 503 (Actual)
Dates: Start 2011-09; Primary Completion 2015-03 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Extent of Implementation of ACP | Year 3
  a. Does the patient have an advance directive or living will or some other written document expressing their wishes? b.patient and/or family been informed of the patients' prognosis? c.Has the patient and/or family been informed about the expected benefits and burdens of various treatment options? d.Has the patient considered how s/he wants to live in the final stages of life and what kinds of medical treatments they would want or not want? e.Have they discussed this with their family? A health care provider? g.Has there been a discussion about their goals of care with their health care provider? If so, are they aware of them? h.Has there been a decision made about medical treatments at the end of life? If so, what role did the patient/family play in that decision-making and was this consistent with their preferred role? i.Is there documentation in the medical record of the overall goals of care?

SECONDARY OUTCOMES:
Effect of an audit and feedback process plus tailored interventions ACP | Year 3
  Compared to baseline, what is the effect of an audit and feedback process coupled with tailored interventions on use of and satisfaction with ACP at the site level?
Impact of ACP on patient/family satisfaction | Year 3
  Compared to those patients who have not undergone an ACP process upon enrolment, what is the impact of ACP on patient/family satisfaction with care, use of life-sustaining technologies, and hospital resources during index hospital admission and long-term health care utilization?
ACP components associated with overall satisfaction | Year 3
  Which components of ACP are more strongly associated with overall satisfaction with EOL communication and decision making?
Comparison of sites with low vs high system level implementation of ACP on satisfaction | Year 3
  At baseline, compared to sites with low degrees of system level implementation, do sites with higher levels of system level integration have a higher prevalence of ACP and greater satisfaction with EOL communication and decision-making?

CONTACTS AND LOCATIONS:
Overall Officials: Daren K Heyland, MD, MSc, Principal Investigator — Queen's University
Locations (9):
- Canada (9):
  - Peter Lougheed Hospital, Calgary, Alberta
  - Foothills Medical Centre, Calgary, Alberta
  - Royal Alexandra Hospital, Edmonton, Alberta
  - Royal Columbian Hospital, New Westminster, British Columbia
  - Vancouver Hospital, Vancouver, British Columbia
  - St Paul's Hospital, Vancouver, British Columbia
  - St.Paul's Hospital, Vancouver, British Columbia
  - Hamilton General Hospital, Hamilton, Ontario
  - Kingston General Hospital, Kingston, Ontario

REFERENCES:
- [Derived] Heyland DK, Heyland R, Dodek P, You JJ, Sinuff T, Hiebert T, Jiang X, Day AG; ACCEPT Study Team and the Canadian Researchers at the End of Life Network (CARENET). Discordance between patients' stated values and treatment preferences for end-of-life care: results of a multicentre survey. BMJ Support Palliat Care. 2017 Sep;7(3):292-299. doi: 10.1136/bmjspcare-2015-001056. Epub 2016 Oct 6. PMID 28827369
- [Derived] Heyland DK, Dodek P, You JJ, Sinuff T, Hiebert T, Tayler C, Jiang X, Simon J, Downar J; ACCEPT Study Team and the Canadian Researchers at the End of Life Network (CARENET). Validation of quality indicators for end-of-life communication: results of a multicentre survey. CMAJ. 2017 Jul 31;189(30):E980-E989. doi: 10.1503/cmaj.160515. PMID 28760834